CLINICAL TRIAL: NCT02201563
Title: A Safety and Feasibility Study of Minocycline Therapy for Management of Adverse Radiation Effects After Brain Metastases Radiosurgery
Brief Title: Minocycline Therapy for Management of Adverse Radiation Effects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Very slow recruitment (only one patient was recruited)
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ajay Niranjan, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14020381
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Irradiation; Adverse Effect
Keywords: Adverse radiation effects (ARE); Radiosurgery; Brain metastases; Minocycline
MeSH Terms: conditions — Brain Neoplasms; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental): oral Minocycline 100 mg twice a day for 3 months.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Oral minocycline (100mg twice a day) for 3 months
  Other Names: Dynacin, Minocin, Minocin PAC, Myrac, Solodyn, Vectrin

SUMMARY:
Stereotactic radiosurgery (SRS) is a well-established treatment for patients with metastatic brain tumors. Although SRS has a very high tumor growth control these interventions are associated with adverse radiation effects (ARE) in approximately 15 % of patients. The traditional approach, and still a mainstay, is the administration of a course of high dose anti-inflammatory corticosteroids. Currently there are no other effective oral neuroprotective agents in clinical practice which can improve outcomes of patients with ARE after radiosurgery for brain metastases.

Minocycline, an antibiotic with a favorable adverse effect profile and pharmacokinetics, has been shown to have neuroprotective properties in experimental models of a variety of neurological diseases, as well as in human clinical trials. The investigators propose a single arm clinical trial, to evaluate the safety and feasibility of minocycline in improving ARE. This study will recruit 15 patients who will be treated with minocycline (100mg BID) for 3 months. This clinical trial has the potential to prove that minocycline therapy is safe in this patient population. In addition, positive results will provide preliminary evidence for its use in an array of radiosurgical indications.

DETAILED DESCRIPTION:
Although stereotactic radiosurgery (SRS) has proven to be highly effective in the management of brain metastases, it is not without risk. Despite selective targeting of lesions and the sharp dose fall-off associated with radiosurgical treatments, adverse radiation effects (AREs) can occur in 10-15% of patients. Adverse radiation effects (AREs) can be defined as unexpected or undesirable post-radiosurgery imaging change regardless of whether it is clinically symptomatic. Patients showing ARE have limited therapeutic options with corticosteroids being the main treatment modality. This single arm clinical trial, will evaluate the safety and feasibility of minocycline in improving AREs. Brain metastases patients with documented AREs will be treated with minocycline (100 mg twice a day) for 3 months in addition to the standard treatment with oral corticosteroids. The investigators anticipate recruiting a total of 15 patients over 12 months.

Primary aim:

The primary aim is of this study to evaluate safety and feasibility of minocycline therapy in patients with ARE after radiosurgery. The investigators' hypothesis is that minocycline will be safe in this patient population. Safety will be assessed by monitoring blood levels of drug, liver enzymes, renal function tests, and monitoring for major and minor side-effects.

Research Strategy The investigators plan to conduct a single arm observational study to evaluate safety and feasibility of minocycline in patients diagnosed with radiosurgery associated adverse radiation effects. In addition to clinical and biochemical monitoring for safety, the investigators will also employ neuroimaging techniques to investigate whether minocycline reduces enhancement at lesion in post contrast T1 weighted MRI and reduces hyper intensity surrounding the tumor as detected by T2 MRI radiosurgery.

Primary Outcomes: 1) The primary clinical outcome will be safety of minocycline use in this patient population.

Secondary outcomes: 1) The investigators will also review brain images in detail to find any evidence of benefit from Minocycline therapy such as reduction or resolution of volume of T2 hyper intensity and contrast enhancement at the lesion (radiation necrosis) at 4-6 weeks and 3 month follow-up. 2) Overall neurological status 3) Change in neurocognitive status, 4) Reduction in the number of patients needing resection 5) Changes in plasma biomarkers, and plasma drug levels.

Target Population: Recruitment will take place at Center of Image-guided Neurosurgery of UPMC. All patients with AREs after brain metastases radiosurgery will be potentially eligible for the study. The investigators anticipate enrolling 15 patients. Patients will be diagnosed based on MRI findings. The investigators will evaluate T1 pre and post contrast, T2, FLAIR and Perfusion MR in order to diagnose ARE. MR spectroscopy or CT Pet will be obtained when clinically indicated. The investigators will use T1/T2 matching and proportion of edema versus lesion volume as a guide for diagnosing ARE.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 90 years
* Males and females.
* Patients must have undergone cranial radiosurgery.
* MRI evidence supporting the diagnosis of ARE and/or surgical biopsy evidence of necrosis without tumor at ≤2 months before study entry.
* Karnofsky performance status of ≥60,
* With or without evidence of progressive neurologic signs or symptoms appropriate to the location of the ARE, and no previous bevacizumab therapy.
* With or without previous chemotherapy for their tumor.
* Routine laboratory study results with bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase and/or alanine aminotransferase <2.5 times the upper limit of normal, creatinine <2.0 times the upper limit of normal.
* Patients with a history of seizures will be required to be receiving anticonvulsant therapy and to be seizure-free for ≥1 week before study.

Exclusion Criteria:

* Significant mass effect requiring resection (as assessed by a clinical neurosurgeon)
* Known hypersensitivity to tetracyclines
* Women of childbearing age must be non-lactating and have a negative urine pregnancy test (adequate birth control includes use of intra uterine device, or a barrier method, e.g. condom, diaphragm). The results of animal studies indicate that tetracyclines cross the placenta and are found in fetal tissues, having potentially toxic effects on the developing fetus (often related to retardation of skeletal development). Evidence of embryo toxicity has been noted in animals treated early in pregnancy. Therefore pregnant women will not be allowed to participate in this study
* Female subjects on oral contraceptives
* Contraindication to undergo MRI
* Significant cardiopulmonary, renal or neurological co-morbidities
* Current diagnosis of major depression, substance abuse, or other psychiatric disorders;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Monitoring for adverse effects of Minocycline | 3 months
  Safety will be assessed by monitoring blood levels of drug, liver enzymes, renal function tests, and monitoring for major and minor side-effects.

SECONDARY OUTCOMES:
Monitoring for imaging improvement | 3 months
  Brain MRIs will be performed to investigate whether minocycline reduces enhancement at lesion in post contrast T1 weighted MRI and reduces hyper intensity surrounding the tumor as detected by T2 MRI radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Niranjan, MD, MBA, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States